CLINICAL TRIAL: NCT01671033
Title: Muscle Relaxation With Biofeedback Via Internet for Panic disorder-a Randomized Pilot Study
Brief Title: Treatment of Panic Disorder Via Internet With a Wireless Temperature Biofeedback Ring
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The drop-out rate was too high.
Sponsor: Chimei Medical Center (Other)
Collaborators: National Cheng Kung University (Other)
Responsible Party: Principal Investigator, Fong-Lin Jang, M.D., Chimei Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB 09902-006
Record Dates: First submitted 2012-08-20; First posted 2012-08-23 (Estimated); Last update posted 2012-08-23 (Estimated); Status verified 2010-04

CONDITIONS: Panic Disorder
Keywords: Panic disorder; cognitive behavior therapy; Internet
MeSH Terms: conditions — Panic Disorder | interventions — Biofeedback, Psychology; Muscle Relaxation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Muscle Relaxation (Experimental): The patients of this arm practice on-line muscle relaxation every day.They complete the Brief Symptom Rating Scale(BSRS), Family APGAR(APGAR), the Chinese-version of the Medical Outcomes Study 36-Item Short Form Health Survey(SF-36), and the panic diary via internet browser. The Panic Disorder Severity Scale(PDSS)and Clinical Global Impression (CGI) were performed by well-trained clinicians.
  Interventions: Behavioral: Muscle Relaxation
- Muscle Relaxation with Biofeedback (Experimental): The patients of this arm practice on-line muscle relaxation with finger temperature biofeedback every day. They complete the Brief Symptom Rating Scale(BSRS), Family APGAR(APGAR), the Chinese-version of the Medical Outcomes Study 36-Item Short Form Health Survey(SF-36), and the panic diary via internet browser. The Panic Disorder Severity Scale(PDSS)and Clinical Global Impression (CGI) were performed by well-trained clinicians.
  Interventions: Behavioral: Biofeedback; Behavioral: Muscle Relaxation
- Waiting-List (No Intervention): The patients of this arm waited for four weeks. They complete the Brief Symptom Rating Scale(BSRS), Family APGAR (APGAR), the Chinese-version of the Medical Outcomes Study 36-Item Short Form Health Survey(SF-36), and the panic diary via internet browser. The Panic Disorder Severity Scale(PDSS)and Impressions-Improvement(CGI) were performed by well-trained clinicians.

INTERVENTIONS:
Behavioral: Biofeedback — Patients with panic disorder practice muscle relaxation with temperature biofeedback monitor, and send the temperature data to server via internet every day. Therapist gives comments and suggestions on line. Patients also have to complete some self-rating scales on browser every day or every week.
  Other Names: finger temperature biofeedback
  Arms: Muscle Relaxation with Biofeedback
Behavioral: Muscle Relaxation — Patients with panic disorder practice muscle relaxation via internet every day. Therapist gives comments and suggestions on line. Patients also have to complete some self-rating scales on browser every day or every week.
  Arms: Muscle Relaxation; Muscle Relaxation with Biofeedback

SUMMARY:
From the scarce literature it showed that computer/internet-aided cognitive behavior therapy (CBT) was superior to waitlist and placebo assignment across outcome measures, and the effects of computer/internet-aided CBT were equal to therapist-delivered treatment across anxiety disorders. The aim of this study is to evidence the effectiveness of internet-based relaxation with biofeedback treatment for panic disorder.

DETAILED DESCRIPTION:
All participants had access to a computer with an internet connection and received the treatment via internet.

ELIGIBILITY:
Inclusion Criteria:

1. The participant must fulfill DSM-IV criteria for panic disorder.
2. The participant must be between 20 and 60 years of age.
3. The participant must have the Panic Disorder Severity Scale(PDSS) score ≧8.
4. If the participant is taking prescribed drugs for panic disorder, a) the dosage have to be constant for 6 weeks before starting treatment, and b) the participant have to agree to keep the dosage constant for 2 months after starting treatment.
5. If the participant was already in therapy, the contact must have lasted at least 3 months and not be based on cognitive behavior therapy.
6. All participants have access to a computer with an Internet connection.

Exclusion Criteria:

1. The participant suffers from any other psychiatric disorder in immediate need of treatment.
2. The participant fulfills DSM-IV criteria for major depression.
3. The participant has epilepsy, kidney problems, strokes, organic brain syndrome, emphysema, heart disorders, or chronic hypertension.
4. The participant has alcoholism or substance dependence.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2010-02; Primary Completion 2010-12 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Score Change of The Panic Disorder Severity Scale(PDSS) | Baseline / Week 4/ Week 8/ Week12/ Week 16

SECONDARY OUTCOMES:
Score Change of relaxation-rating | Baseline / Week 4/ Week 8/ Week 12/ Week 16

CONTACTS AND LOCATIONS:
Overall Officials: Fong-Lin Jang, M.D., Study Director — Chimei Medical Center
Locations (1):
- Chimei Medical Center, Tainan, Taiwan